CLINICAL TRIAL: NCT03870815
Title: Registry for Long-term Clinical Outcomes and Prognostic Factors in Patient With Coronary Artery Disease Undergoing Coronary Artery Bypass Graft Surgery or Percutaneous Coronary Intervention With Second Generation Drug-Eluting Stent
Brief Title: Long-term Outcomes and Prognostic Factors in Patient Undergoing CABG or PCI
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Young Bin Song, Associate Professor, Samsung Medical Center
Other Study IDs: CABG2019
Record Dates: First submitted 2019-03-10; First posted 2019-03-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Ischemic Heart Disease
Keywords: Ischemic heart disease; Coronary artery bypass grafting; Percutaneous coronary intervention
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CABG: Patients with CAD who undergoing CABG
  Interventions: Procedure: CABG
- PCI: Patients with CAD who undergoing PCI with DES
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: CABG — Patients who undergoing CABG
  Groups: CABG
Procedure: PCI — Patients who undergoing PCI with DES
  Groups: PCI

SUMMARY:
1. To evaluate the long-term clinical outcomes and prognostic factors in patients with coronary artery disease undergoing coronary artery bypass graft surgery.
2. To evaluate the long-term clinical outcomes and prognostic factors in patients with coronary artery disease undergoing percutaneous coronary intervention with drug-eluting stent.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) still remains one of the world's leading causes of death, despite markedly improvement of devices and technologies on past several decades. The treatment strategy for CAD included medical treatment, percutaneous coronary intervention (PCI), and coronary-artery bypass grafting (CABG). CABG is a procedure in which autologous arteries or veins are used as grafts to bypass coronary arteries that are partially or completely obstructed by atherosclerotic plaque. During the past decade, there has been nearly a 30% decline in CABG procedures, despite abundant evidence to support the effectiveness and safety of the operation.This decline has been accompanied by a corresponding increase in PCI. To date, there have been numerous studies to compare the clinical outcomes between PCI and CABG for patients with CAD. Among them, SYNTAX (Synergy between PCI with Taxus and Cardiac Surgery) trial demonstrated CABG is associated with lower incidence of major adverse cardiac and cerebrovascualr events in patients with high SYNTAX score, compared with PCI. In this regard, the current guidelines recommend that CABG is preferred method for care of stable ischemic heart disease patients with three-vessel or left main coronary artery disease. However, most randomized controlled studies do not reflect the contemporary practice, because they have been performed in the era of bare metal stents or first-generation drug-eluting stent (DES). In addition, there have been limited data regarding the prognostic factors for long-term clinical outcomes in patients undergoing PCI with DES or CABG. Therefore, the investigators sought to compare the clinical outcomes between PCI with DES or CABG, and to identify prognostic factors for long-term clinical outcomes in patients who underwent PCI with DES or CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suspected ischemic heart disease and underwent CABG or PCI with DES

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 10,000 patients with suspected ischemic heart disease and who underwent PCI with DES or CABG.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Cardiac Death | 5-Year after the index procedure
  death from cardiac-cause

SECONDARY OUTCOMES:
All-cause Death | 5-Year after the index procedure
  death from any-cause
Myocardial infarction | 5-Year after the index procedure
  Myocardial infarction without peri-procedural myocardial infarction
Target-vessel revascularization | 5-Year after the index procedure
  ischemia-driven or all
Any revascularization | 5-Year after the index procedure
  ischemia-driven or all
Bleeding | 5-Year after the index procedure
  BARC type 2-5
Cerebrovascular accident | 5-Year after the index procedure
  Ischemic or hemorrhagic
MACCE (major adverse cardiac and cerebrovascular accident) | 5-Year after the index procedure
  a composite of death, myocardial infarction, and cerebrovascular accident

CONTACTS AND LOCATIONS:
Overall Officials: Young Bin Song, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee SY, Cho YH, Sung K, Kim WS, Lee SJ, Kwon W, Lee JY, Lee SH, Shin D, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Choi KH, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Jeong DS, Lee JM. Intravascular Imaging-Guided PCI vs Coronary Artery Bypass Grafting for Left Main or 3-Vessel Disease. JACC Cardiovasc Interv. 2025 Sep 8;18(17):2077-2088. doi: 10.1016/j.jcin.2025.06.034. Epub 2025 Aug 27. PMID 40864021
- [Derived] Lee SY, Lee SJ, Kwon W, Lee SH, Shin D, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Choi KH, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Lee JY, Lee JM, Investigators TR. Outcomes of intravascular imaging-guided percutaneous coronary intervention according to lesion complexity. EuroIntervention. 2025 Feb 3;21(3):e171-e182. doi: 10.4244/EIJ-D-24-00755. PMID 39901632
- [Derived] Lee SH, Jo J, Yang JH, Kim SM, Choi KH, Song YB, Jeong DS, Lee JM, Park TK, Hahn JY, Choi SH, Chung SR, Cho YH, Sung K, Kim WS, Gwon HC, Lee YT. Clinical Impact of Sarcopenia Screening on Long-Term Mortality in Patients Undergoing Coronary Bypass Grafting. J Cachexia Sarcopenia Muscle. 2024 Dec;15(6):2842-2851. doi: 10.1002/jcsm.13645. Epub 2024 Nov 8. PMID 39513369
- [Derived] Joh HS, Kwon W, Shin D, Lee SH, Hong YJ, Hong D, Lee SY, Park H, Kim S, Lee SY, Koh JS, Kim H, Kim CJ, Choo EH, Yoon HJ, Park SD, Jeon KH, Bae JW, Ahn SG, Kim SE, Choi KH, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Gwon HC, Lee JM. Drug-Coated Balloon Angioplasty in Patients Undergoing Complex Percutaneous Coronary Intervention. JACC Asia. 2024 Jun 18;4(7):519-531. doi: 10.1016/j.jacasi.2024.04.007. eCollection 2024 Jul. PMID 39101114
- [Derived] Kwon W, Hong D, Choi KH, Lee SH, Shin D, Lee JY, Lee SJ, Lee SY, Kim SM, Yun KH, Cho JY, Kim CJ, Ahn HS, Nam CW, Yoon HJ, Park YH, Lee WS, Park TK, Yang JH, Choi SH, Gwon HC, Song YB, Hahn JY, Lee JM; RENOVATE-COMPLEX-PCI Investigators. Intravascular Imaging-Guided Percutaneous Coronary Intervention Before and After Standardized Optimization Protocols. JACC Cardiovasc Interv. 2024 Jan 22;17(2):292-303. doi: 10.1016/j.jcin.2023.10.062. PMID 38267144
- [Derived] Jang WJ, Choi KH, Kim J, Yang JH, Hahn JY, Choi SH, Gwon HC, Cho YH, Sung K, Kim WS, Jeong DS, Song YB. Impact of gender on mid-term prognosis of patients undergoing coronary artery bypass grafting. PLoS One. 2023 Mar 2;18(3):e0279030. doi: 10.1371/journal.pone.0279030. eCollection 2023. PMID 36862681
- [Derived] Kwon W, Choi KH, Jeong DS, Lee SY, Lee JM, Park TK, Yang JH, Hahn JY, Choi SH, Chung SR, Cho YH, Sung K, Kim WS, Gwon HC, Lee YT, Song YB. Comparison of long-term cardiovascular and renal outcomes between percutaneous coronary intervention and coronary artery bypass grafting in multi-vessel disease with chronic kidney disease. Front Cardiovasc Med. 2022 Sep 12;9:951113. doi: 10.3389/fcvm.2022.951113. eCollection 2022. PMID 36172577
- [Derived] Choi KH, Song YB, Jeong DS, Jang YH, Hong D, Lee SY, Youn T, Bak M, Min KM, Lee JM, Park TK, Yang JH, Hahn JY, Choi JH, Choi SH, Chung SR, Cho YH, Sung K, Kim WS, Gwon HC, Lee YT. Differential effects of dual antiplatelet therapy in patients presented with acute coronary syndrome vs. stable ischaemic heart disease after coronary artery bypass grafting. Eur Heart J Cardiovasc Pharmacother. 2021 Nov 3;7(6):517-526. doi: 10.1093/ehjcvp/pvaa080. PMID 33075126